CLINICAL TRIAL: NCT06758063
Title: Impact of Physical Activities on Balance in Patient With Post-surgical Strabismic Amblyopia
Brief Title: Impact of Physical Activities on Balance in Patient With Strabismic Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amany Refaat Mohamed Abdel Wahid (Other)
Responsible Party: Sponsor-Investigator, Amany Refaat Mohamed Abdel Wahid, Lecturer at department of Surgery, faculty of Physical Therapy, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.R/012/005408
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Balance Control
Keywords: Balance; stabismus; amblyopia; physical therapy; exercises
MeSH Terms: conditions — Amblyopia; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise therapy (Other): this group will apply balance exercises two times a week for three months
  Interventions: Other: exercises therapy
- traditional eye care (No Intervention): This group will receive traditional eye observation post strabismus surgery

INTERVENTIONS:
Other: exercises therapy — exercises to improve balance of the body
  Arms: exercise therapy

SUMMARY:
The aim of this study is to determine the effect of physical activities on balance in patient with amblyopia after strabismus surgery. Patients with strabismus have more difficulty in maintaining postural control in the presence of misleading signals. Through this study the patients will apply physical therapy sessions to improve balance for strabismic amblyopic patient post-surgery.

DETAILED DESCRIPTION:
* Patients will be informed about measurement and treatment procedure, also about the effect of physical activity on improving balance post strabismus surgery.
* Patients will be asked to follow physician instructions.
* Patients will be asked to avoid participation in any rehabilitation program prior to the study which may affect the result of the study.
* Measurement procedures will be applied for each patient.
* The therapeutic group will receive 2 sessions per week for 12 weeks. The duration of each session is 45 min.
* They will start the treatment program after 2 months of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients received strabismus operation.
* Patients are suffering from balance problem due to strabismus
* Patients are suffering from strabismus amblyopia
* They will be selected from Outpatient Clinic of Research Institute of Ophthalmology.
* Patients will begin the training program after 2 months of operation.
* Patient with intermittent exotropia

Exclusion Criteria:

* - Patients with a diagnosis of vestibular, neurological and psychiatric diseases
* Moderate and severe amblyopia,
* Any disease that can cause imbalance syndrome or limitation of movement
* A history of falling without a cause in the last 6 months and
* Using drugs affecting the central nervous system
* Patient who didn't complete the physiotherapy training program for 3 months.
* Muscular disorders that will impair performance during training.
* Any organic lesion in the eye.
* Malignant conditions.
* Children who can't understand the therapist's instructions and orders
* Amblyopia which is not related to strabismus condition

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
The Berg Balance Scale | From enrollment to the end of treatment at 12 weeks
  * The scale involves 14 mobility tasks, with the tasks varying in degrees of difficulty. The tasks are divided into 3 domains: sitting balance, standing balance, and dynamic balance.
  * Each task is graded on a 5-point ordinal scale that ranges from 0 to 4 for a maximum score of 56. In general, a score of 0 is given when the individual is unable to perform the task, and a score of 4 is given when able to complete the given task independently
Dynamic single leg stance test | From enrollment to the end of treatment at 12 weeks
  1. The subject begins in quiet standing with hands on the hips.
  2. The subject lifts one leg off the ground and stands unassisted.
  3. Time starts when the foot is lifted off the ground
  4. Time stops when the lifted foot either makes contact with the ground, makes contact with the stance limb, when the stance foot moves laterally on the floor, or when the hands leave the hips.
  5. Dynamic posture tasks will applied during the test

CONTACTS AND LOCATIONS:
Overall Officials: Amany R M Abdel Wahid, Doctoral degree, Principal Investigator — Lecturer at faculty of physical therapy, Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Giza Governorate, Egypt